CLINICAL TRIAL: NCT05239104
Title: Laos Out-Of-Pocket Costs: an Observational Study on the Impact of Severe Childhood Illness on the Health, Wealth and Wellbeing of Household Members in Lao People's Democratic Republic
Brief Title: Laos Out-Of-Pocket Costs: an Observational Study on the Impact of Severe Childhood Illness on the Health, Wealth and Wellbeing of Household Members in Laos
Acronym: LOOP
Status: Completed | Type: Observational
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: 81864
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Health Care Economics; Child Health; Cost of Illness; Burden of Illness
Keywords: health behaviour; health equity; poverty; hospital costs; developing countries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children aged 1 month - 14 years 11 months with a severe illness/injury: Children aged 1 month - 14 years 11 months presenting to hospital with symptoms of an acute "severe" illness/injury that started within the last 2 weeks. "Severe" defined as a child showing emergency signs or requiring hospital admission for treatment.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study with no intervention

SUMMARY:
This will be a prospective longitudinal study of children attending hospital for treatment of a severe illness with community follow-up in Lao People's Democratic Republic (Lao PDR). The study aims to summarise and describe short-term health and economic impacts of a severe childhood illness requiring hospital admission, from a household perspective.

DETAILED DESCRIPTION:
This study aims to measure the out-of-pocket (OOP) expenses for households related to a severe acute illness/injury in children under five years presenting to hospitals in Lao PDR. Financial protection will be measured by determining proportions of households led to catastrophic health expenditures and impoverishment from OOP expenses, with further equity analyses across wealth quintiles, geographical residence, sex, parental education and ethnic subpopulations. Physical health and mental wellbeing outcomes of participants and household members will also be assessed to determine the multifaceted impact of severe childhood disease on a household.

Participants will be recruited in outpatients, the emergency department (ED) or during hospital admission. Information on the participant's illness will be collected through health records where available. Household demographic data, financial costs and coping strategies associated with illness and health/wellbeing outcomes will be collected through parent/caregiver structured questionnaires. These will be conducted during presentation to outpatients/ED or during admission on the wards, with follow-up at 2 weeks and at 2 months post-presentation or post-discharge.

Average total household out-of-pocket (OOP) expenses associated with the illness will be presented for the study population. An equity analysis will be performed by disaggregating and comparing mean/median OOP costs across wealth quintiles, sex, geographical location, parental education and ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* Child is aged between 1 month -14 years 11 months at the time of admission/presentation to outpatient / ED / hospital
* Child presents to or is admitted to hospital at one of the participating study site hospitals within the time period of the study
* Child presents with symptoms of acute illness that started within the last 2 weeks (14 days) prior to hospital presentation. This will include children with a chronic illness but with new onset of symptoms within last 2 weeks.
* Child is assessed by a health officer at the participating study site hospital and is deemed to have a "severe" illness/injury. A "severe" illness/injury will be defined as a child showing any emergency signs as outlined in the WHO Pocketbook, second edition:

OR Requires hospital admission/transfer to another health facility for further investigations and/or treatment for their acute illness/injury that cannot be performed in an outpatient setting or ED. This may include but is not limited to: transfer to another hospital with intensive care unit (ICU), intravenous (IV) medication or fluids; enteral nutrition; oxygen therapy; surgery.

• Parent/guardian has provided written informed consent, and will be available for the duration of the study follow-up period.

Exclusion Criteria:

* Child <1 month or >14 years 11 months at time of presentation to hospital
* Child with symptoms that started >2 weeks (>14 days) prior to hospital presentation
* Child admitted to the neonatal intensive care unit (NICU)
* Child admitted to hospital for a planned procedure or planned treatment of a chronic medical condition (eg. Tonsillectomy, replacement of ventriculoperitoneal shunt or percutaneous endoscopic gastronomy (PEG) tube, tune up for cystic fibrosis, chemotherapy, palliative care),
* Child already enrolled into this study from a previous hospital admission
* Child discharged prior to screening and informed consent processes by study team members.

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 1 month - 14 years 11 months with a "severe" illness/injury who is admitted or presented to outpatient/ED/ward at one of the participating study site hospitals in Lao PDR.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Mean total out-of-pocket (OOP) expenses | 2 months
  Total OOP expenses are the combined total of direct (medical and non-medical) OOP expenses and indirect costs per household.
  Data will be collected from a parent/guardian questionnaire developed for the study and expenses will be calculated from onset of symptoms up to 2 months post-discharge from hospital; presented in Lao kip (LAK) and US dollars (USD). Outcome will be presented as mean total OOP expenses per household.
  Direct medical OOP costs include: consultation fees, fees for diagnostics, medicine and other treatment/remedy costs, hospital bed fees, transfer costs, insurance co-pay if applicable.
  Direct non-medical OOP costs include: travel costs for patient and accompanying carer/household member/s, daily living expenses for patient and accompanying carer/household member/s including food, childcare costs for other children at home, lodging.
  Indirect costs include: travel time, loss of income incurred from the cessation or reduction of work productivity.

SECONDARY OUTCOMES:
Total number and percentage of households experiencing Catastrophic Health Expenditure (CHE) set at 10% total annual household expenditure (CHE10a) | 2 months
  CHE: defined as when the total OOP expenses exceeds a threshold proportion of household expenditures.
  CHE10a: The primary CHE threshold will be set at 10% of total annual household expenditure to align with Sustainable Development Goal (SDG) indicator 3.8.2.
  OOP expenses and household expenditures will be collected through a study developed questionnaire and CHE10a will be presented as a total number and as a percentage of study participants.
Total number and percentage of households experiencing CHE set at 10% monthly household expenditure (CHE10m) | 2 months
  CHE10m: a secondary CHE threshold will be set at 10% of monthly household expenditure to show the immediate financial impact of the illness OOP expenses and household expenditures will be collected through a study developed questionnaire and CHE10m will be presented as a total number and as a percentage of study participants.
Total number and percentage of households experiencing CHE set at 40% annual capacity to pay (CHE40a) | 2 months
  CHE40a: a secondary CHE threshold will be set at 40% annual capacity to pay (CTP) with previous studies suggesting it more effective at identifying poorer households.
  CTP: defined as the total household expenditures minus necessary subsistence expenditures (food, housing, utilities).
  OOP expenses and household expenditures will be collected through a study developed questionnaire and CHE40a will be presented as a total number and as a percentage of study participants.
Total number and percentage of households experiencing CHE set at 40% monthly CTP (CHE40m) | 2 months
  CHE40m: a secondary CHE threshold will be set at 40% monthly CTP with previous studies suggesting it more effective at identifying poorer households.
  CTP: defined as the total household expenditures minus necessary subsistence expenditures (food, housing, utilities).
  OOP expenses and household expenditures will be collected through a study developed questionnaire and CHE40m will be presented as a total number and as a percentage of study participants.
Total number and percentage of households experiencing Impoverishment Health Expenditure (IHE) set at international poverty line (IHE-i) | 2 months
  IHE: defined as households that fall below the poverty line due to the OOP payments associated with the severe illness.
  IHE-i: primary threshold will be presented for the international poverty line (US$1.90 per person per day) to align with SDG target 1.1.
  OOP expenses will be collected through a study developed questionnaire and IHE-i will be presented as a total number and as a percentage of study participants.
Total number and percentage of households experiencing Impoverishment Health Expenditure (IHE) set at national poverty line (IHE-n) | 2 months
  IHE-n: a secondary threshold will be presented for the national poverty line (LAK 280,910 per person per month) OOP expenses will be collected through a study developed questionnaire and IHE-n will be presented as a total number and as a percentage of study participants.
Median number of coping strategies used by households | 2 months
  Strategies households employ to finance the OOP costs related to the severe illness, defined as: use of savings, borrowing, help from others, asset sales, delayed plans, and/or reduced consumption.
  Data will be collected through a study developed questionnaire and will be presented as median number of coping strategies used per household.
Health outcomes of participating children - mean length of hospital admission | 2 months
  Length of hospital admission measured in days Data will be collected from participants' hospital medical records and will be presented as mean length of hospital admission per participant.
Health outcome of participating children - total number and percentage of deaths | 2 months
  Total number of deaths of participating children during study period, presented as total number and percentage of study population.
  Data will be collected from parent/guardian report in study developed questionnaire
Health outcome of participating children - total number and percentage of participating children reporting each recovery status | at 2 weeks post-discharge from hospital
  Recovery status defined as level of recovery from serious illness as reported by parent/guardian (full recovery, partial recovery, sicker than when left hospital, death). Recovery status will be presented as total number and percentage of study population reporting each recovery status and then ranked from highest to lowest percentage. Data will be collected from a study developed questionnaire
Health outcome of participating children - total number and percentage of participating children reporting each recovery status | at 2 months post-discharge from hospital
  Recovery status defined as level of recovery from serious illness as reported by parent/guardian (full recovery, partial recovery, sicker than when left hospital, death). Recovery status will be presented as total number and percentage of study population reporting each recovery status and then ranked from highest to lowest percentage. Data will be collected from a study developed questionnaire
Health outcome of participating children - total number of children returning to ED/hospital | 2 months
  Total number of participating children returning to ED/hospital as a complication of the initial severe illness.
  Data will be collected from parent/guardian report in study developed questionnaire and will be presented as total number and as percentage of study population.
Health outcome of participating children - mean change in nutritional status | 2 months
  Change in nutritional status defined as change in weight-for-height score presented as standard deviation (or z-score) from outpatient/ED presentation or hospital discharge. The z-score are compared to reference population z-scores as defined in WHO global database growth charts.
  Data will be collected through anthropometry measures (height and weight) and will be presented as mean difference in z-score for study population from start to end of study period.
Health outcome of participating children - total number and percentage with moderate to severe wasting | At enrolment (day 0)
  Number of participants with wasting defined as weight-for-height score presented as standard deviation <-2 (z-score <-2).
  Data will be collected through anthropometry measures (height and weight) and will be presented as total number and as percentage of study population.
Health outcome of participating children - total number and percentage with moderate to severe wasting | 2 months
  Number of participants with wasting defined as weight-for-height z-score <-2. Data will be collected through anthropometry measures (height and weight) and will be presented as total number and as percentage of study population.
Health outcome of participating children - total number and percentage of children not admitted to hospital or early discharge from hospital | 2 months
  Total number of participants with patient/caregiver decision to not be admitted to hospital from outpatients/ED or discharge early from hospital against medical advice.
  Data will be collected from parent/guardian report in study developed questionnaire or participants' hospital medical records and will be presented as total number as percentage of study population.
Health and wellbeing outcomes of participant household members - median number of household members with same illness as participant child | 2 months
  Number of household members with same illness as participant. Data will be collected from parent/guardian report in study developed questionnaire and presented as median number of sick household members per household.
Health and wellbeing outcomes of participant household members - median number of deaths | 2 months
  Number of deaths of household members within each household during study period.
  Data will be collected from parent/guardian report in study developed questionnaire and presented as median number of deaths of household members per household.
Health and wellbeing outcomes of primary caregivers - total number and percentage of primary caregivers with worse nutritional status | 2 months
  Primary caregivers with worse nutritional status, defined as unintentional weight loss of >5% from recruitment stage; and/or primary caregivers that are pushed into category of underweight (BMI < 18 kg/m2) from recruitment stage.
  Data will be collected from anthropometry measures (height and weight) of primary caregivers and will be presented as total number and as a percentage of primary caregivers.
Health and wellbeing outcomes of primary caregiver - mean change in quality of life score (physical health) | 2 months
  The WHO Quality of Life - abbreviated version tool (WHOQOL-BREF) is a short-version of the WHOQOL-100, a validated tool developed by WHO to assess quality of life. The WHOQOL-BREF is a 26-item questionnaire assessing four domains contributing to quality of life (physical health, psychological health, social relationships, environment). Each domain will produce a score from 0-100, with a higher score indicating a higher quality of life for that domain.
  The WHOQOL-BREF questionnaire will be conducted with the primary caregiver. Score for the physical health domain will be presented as mean difference in scores from start to end of study period.
Health and wellbeing outcomes of primary caregiver - mean change in quality of life score (psychological health) | 2 months
  The WHO Quality of Life - abbreviated version tool (WHOQOL-BREF) is a short-version of the WHOQOL-100, a validated tool developed by WHO to assess quality of life. The WHOQOL-BREF is a 26-item questionnaire assessing four domains contributing to quality of life (physical health, psychological health, social relationships, environment). Each domain will produce a score from 0-100, with a higher score indicating a higher quality of life for that domain.
  The WHOQOL-BREF questionnaire will be conducted with the primary caregiver. Score for the psychological health domain will be presented as mean difference in scores from start to end of study period.
Health and wellbeing outcomes of primary caregiver - mean change in quality of life score (social relationships) | 2 months
  The WHO Quality of Life - abbreviated version tool (WHOQOL-BREF) is a short-version of the WHOQOL-100, a validated tool developed by WHO to assess quality of life. The WHOQOL-BREF is a 26-item questionnaire assessing four domains contributing to quality of life (physical health, psychological health, social relationships, environment). Each domain will produce a score from 0-100, with a higher score indicating a higher quality of life for that domain.
  The WHOQOL-BREF questionnaire will be conducted with the primary caregiver. Score for the social relationships domain will be presented as mean difference in scores from start to end of study period.
Health and wellbeing outcomes of primary caregiver - mean change in quality of life score (environment) | 2 months
  The WHO Quality of Life - abbreviated version tool (WHOQOL-BREF) is a short-version of the WHOQOL-100, a validated tool developed by WHO to assess quality of life. The WHOQOL-BREF is a 26-item questionnaire assessing four domains contributing to quality of life (physical health, psychological health, social relationships, environment). Each domain will produce a score from 0-100, with a higher score indicating a higher quality of life for that domain.
  The WHOQOL-BREF questionnaire will be conducted with the primary caregiver. Score for the environment domain will be presented as mean difference in scores from start to end of study period.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Russell, BMBS FRACP MPHTM PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Lao-Oxford-Mahosot-Hospital Wellcome Trust Research Unit (LOMWRU), Vientiane, Laos

IPD SHARING:
Plan to Share IPD: Yes
Beginning 0 (zero) months following analysis and article publication, individual participant data (IPD) will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access.
  • Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures, and appendices) will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will be available from date summary data is published
Access Criteria: Requests to access IPD are to be made with the principal investigator who will review requests and share IPD with supporting information as ethically appropriate. All IPD will be de-identified

REFERENCES:
- [Background] Zhang S, Sammon PM, King I, Andrade AL, Toscano CM, Araujo SN, Sinha A, Madhi SA, Khandaker G, Yin JK, Booy R, Huda TM, Rahman QS, El Arifeen S, Gentile A, Giglio N, Bhuiyan MU, Sturm-Ramirez K, Gessner BD, Nadjib M, Carosone-Link PJ, Simoes EA, Child JA, Ahmed I, Bhutta ZA, Soofi SB, Khan RJ, Campbell H, Nair H. Cost of management of severe pneumonia in young children: systematic analysis. J Glob Health. 2016 Jun;6(1):010408. doi: 10.7189/jogh.06.010408. PMID 27231544
- [Background] Barennes H, Frichittavong A, Gripenberg M, Koffi P. Evidence of High Out of Pocket Spending for HIV Care Leading to Catastrophic Expenditure for Affected Patients in Lao People's Democratic Republic. PLoS One. 2015 Sep 1;10(9):e0136664. doi: 10.1371/journal.pone.0136664. eCollection 2015. PMID 26327558
- [Background] Wagstaff A, Flores G, Hsu J, Smitz MF, Chepynoga K, Buisman LR, van Wilgenburg K, Eozenou P. Progress on catastrophic health spending in 133 countries: a retrospective observational study. Lancet Glob Health. 2018 Feb;6(2):e169-e179. doi: 10.1016/S2214-109X(17)30429-1. Epub 2017 Dec 13. PMID 29248367
- [Background] Xu K, Evans DB, Kawabata K, Zeramdini R, Klavus J, Murray CJ. Household catastrophic health expenditure: a multicountry analysis. Lancet. 2003 Jul 12;362(9378):111-7. doi: 10.1016/S0140-6736(03)13861-5. PMID 12867110
- [Background] Xu K, Evans DB, Carrin G, Aguilar-Rivera AM, Musgrove P, Evans T. Protecting households from catastrophic health spending. Health Aff (Millwood). 2007 Jul-Aug;26(4):972-83. doi: 10.1377/hlthaff.26.4.972. PMID 17630440
- [Background] Grepin KA, Irwin BR, Sas Trakinsky B. On the Measurement of Financial Protection: An Assessment of the Usefulness of the Catastrophic Health Expenditure Indicator to Monitor Progress Towards Universal Health Coverage. Health Syst Reform. 2020 Dec 1;6(1):e1744988. doi: 10.1080/23288604.2020.1744988. PMID 33416439
- [Background] Memirie ST, Metaferia ZS, Norheim OF, Levin CE, Verguet S, Johansson KA. Household expenditures on pneumonia and diarrhoea treatment in Ethiopia: a facility-based study. BMJ Glob Health. 2017 Jan 18;2(1):e000166. doi: 10.1136/bmjgh-2016-000166. eCollection 2017. PMID 28589003
- [Background] Wagstaff A, Flores G, Smitz MF, Hsu J, Chepynoga K, Eozenou P. Progress on impoverishing health spending in 122 countries: a retrospective observational study. Lancet Glob Health. 2018 Feb;6(2):e180-e192. doi: 10.1016/S2214-109X(17)30486-2. Epub 2017 Dec 13. PMID 29248366
- [Background] Wagstaff A, Lindelow M. Are health shocks different? Evidence from a multishock survey in Laos. Health Econ. 2014 Jun;23(6):706-18. doi: 10.1002/hec.2944. Epub 2013 Jun 13. PMID 23765700
- [Background] Hogan DR, Stevens GA, Hosseinpoor AR, Boerma T. Monitoring universal health coverage within the Sustainable Development Goals: development and baseline data for an index of essential health services. Lancet Glob Health. 2018 Feb;6(2):e152-e168. doi: 10.1016/S2214-109X(17)30472-2. Epub 2017 Dec 13. PMID 29248365
- [Background] Alam K, Mahal A. Economic impacts of health shocks on households in low and middle income countries: a review of the literature. Global Health. 2014 Apr 3;10:21. doi: 10.1186/1744-8603-10-21. PMID 24708831
- [Background] Bodhisane S, Pongpanich S. The impact of National Health Insurance upon accessibility of health services and financial protection from catastrophic health expenditure: a case study of Savannakhet province, the Lao People's Democratic Republic. Health Res Policy Syst. 2019 Dec 16;17(1):99. doi: 10.1186/s12961-019-0493-3. PMID 31842882
- [Background] Barasa EW, Ayieko P, Cleary S, English M. Out-of-pocket costs for paediatric admissions in district hospitals in Kenya. Trop Med Int Health. 2012 Aug;17(8):958-61. doi: 10.1111/j.1365-3156.2012.03029.x. Epub 2012 Jun 21. PMID 22716184
- [Background] Sultana M, Alam NH, Ali N, Faruque ASG, Fuchs GJ, Gyr N, Chisti MJ, Ahmed T, Gold L. Household economic burden of childhood severe pneumonia in Bangladesh: a cost-of-illness study. Arch Dis Child. 2021 Jun;106(6):539-546. doi: 10.1136/archdischild-2020-320834. Epub 2021 Apr 27. PMID 33906852
- [Background] Alamgir NI, Naheed A, Luby SP. Coping strategies for financial burdens in families with childhood pneumonia in Bangladesh. BMC Public Health. 2010 Oct 19;10:622. doi: 10.1186/1471-2458-10-622. PMID 20955627
- [Background] Gray AZ, Morpeth M, Duke T, Peel D, Winter C, Satvady M, Sisouk K, Prasithideth B, Detleuxay K. Improved oxygen systems in district hospitals in Lao PDR: a prospective field trial of the impact on outcomes for childhood pneumonia and equipment sustainability. BMJ Paediatr Open. 2017 Aug 31;1(1):e000083. doi: 10.1136/bmjpo-2017-000083. eCollection 2017. PMID 29637121
- [Background] Cederholm T, Bosaeus I, Barazzoni R, Bauer J, Van Gossum A, Klek S, Muscaritoli M, Nyulasi I, Ockenga J, Schneider SM, de van der Schueren MA, Singer P. Diagnostic criteria for malnutrition - An ESPEN Consensus Statement. Clin Nutr. 2015 Jun;34(3):335-40. doi: 10.1016/j.clnu.2015.03.001. Epub 2015 Mar 9. PMID 25799486